CLINICAL TRIAL: NCT06493188
Title: Effectiveness of Low-fidelity Versus High-fidelity Interprofessional Simulation on the Acquisition of Theoretical and Practical Knowledge of Arterial Blood Gas Testing: a Parallel Randomized Controlled Trial
Brief Title: Low VS High-fidelity Interprofessional Simulation for ABG Skills Acquisition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Fondazione CRT, Torino (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INTSIM_GB_UNITO_01
Record Dates: First submitted 2024-06-27; First posted 2024-07-09 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Interprofessional Relations; Self Efficacy; Knowledge, Attitudes, Practice
Keywords: Interprofessional education; Simulation; Arterial Blood Gas test; Self-efficacy; Knowledge acquisition
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - High-fidelity interprofessional simulation (Experimental): The interprofessional simulation activity will be conducted in the immersive medical training room. ABG will be performed on a arm simulator. The patient will be personified by an actor with a medical background following a script. A maximum of 10 minutes will be given to address each case.
  Interventions: Other: High-fidelity interprofessional simulation
- Control Group - Low-fidelity interprofessional simulation (Active Comparator): This interprofessional simulation activity will be conducted in a room that will be equipped with tables and chairs. The same clinical cases will be provided using printed documents and clinical charts. A time of 10 minutes will be given to address each case.
  Interventions: Other: Low-fidelity interprofessional simulation

INTERVENTIONS:
Other: High-fidelity interprofessional simulation — Students will participate in realistic (high-fidelity) interprofessional simulation scenarios to practice and interpret ABG procedures.
  Arms: Intervention Group - High-fidelity interprofessional simulation
Other: Low-fidelity interprofessional simulation — Students will take part in low-fidelity interprofessional simulation scenarios. Cases will be discussed, and reflection on ABG execution and interpretation will be guided using paper descriptions and clinical files.
  Arms: Control Group - Low-fidelity interprofessional simulation

SUMMARY:
This randomized clinical trial will evaluate the effectiveness of an interprofessional simulation intervention for medical and nursing students.

The primary aim is to compare the effectiveness of high-fidelity versus low-fidelity interprofessional simulation in improving knowledge and skills related to the ABG test. The hypothesis is that participants in the high-fidelity interprofessional simulation group will develop better knowledge and skills for ABG testing compared to those in the low-fidelity group.

The secondary aims are to evaluate the effectiveness of high-fidelity interprofessional simulation compared to low-fidelity interprofessional simulation in (i) enhancing self-efficacy and self-confidence in learning, and (ii) improving interprofessional education and satisfaction with the simulation experience. It is hypothesized that participants in the high-fidelity interprofessional simulation group will report higher levels of self-efficacy, self-confidence, interprofessional education, and satisfaction with the learning experience post-intervention compared to those in the low-fidelity interprofessional simulation group.

The key questions it seeks to address are:

1. Does high-fidelity interprofessional simulation help in developing better technical skills for ABG testing?
2. Does high-fidelity interprofessional simulation lead to greater self-efficacy and self-confidence?
3. Does high-fidelity interprofessional simulation lead to greater satisfaction with the experience, readiness for interprofessional simulation, and better perceptions of interprofessional education?

The researchers will compare high-fidelity interprofessional simulation (immersive medical training room with an actor) to low-fidelity interprofessional simulation (a structured clinical case analysis) to assess whether high-fidelity simulation effectively enhances knowledge and skills on arterial blood gas tests, as well as interprofessional collaboration and attitudes.

Participants will:

* Attend brief interactive lessons on the principles, technique, and interpretation of arterial blood gas tests.
* Participate in a series of clinical-based interprofessional simulation scenarios delivered in low- or high-fidelity.

DETAILED DESCRIPTION:
After randomization, participants will be assigned sequentially into ten groups to form five high-fidelity interprofessional simulation groups and five low-fidelity interprofessional simulation groups. Each group will consist of six students, including three medical students and three nursing students.

Students will be asked to review and sign the informed consent form to confirm their participation in the study.

Participants will be asked to complete the baseline assessment by completing a questionnaire set. They will be subjected to a brief educational video covering the definition and purpose of the ABG test, the diagnostic and clinical rationale for conducting it, and the technique, including patient assessment, required equipment, factors to consider before performing the procedure, questions to ask the patient, identification of the puncture site, sampling steps, and proper disposal of materials. Additionally, a brief interpretation of ABG test results will be provided, focusing on pH values, carbon dioxide levels, and bicarbonate levels to identify the four main diagnoses: respiratory acidosis, metabolic acidosis, respiratory alkalosis, and metabolic alkalosis.

At the end of the video presentation, participants will be informed about which group they have been assigned to.

During the simulation activities, two independent observers will assess the performance of participants.

At the end of the simulation activities, all students from both groups will be taken separately to designated plenary rooms, where a member of the research team will conduct a debriefing session.

At the conclusion of the debriefing session, each participant will be asked to complete a set of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Early-career students (First-year Nursing Bachelor's Degree; second-year Medicine & Surgery Degree)
* Regularly enrolled in their courses (attended at least 70% of classes)
* Proficient in English (reading and speaking)
* Aged 18 years or older

Exclusion Criteria:

* Students who have previously taken classes on arterial blood gas sampling
* Those who have prior work experience as healthcare professionals (e.g., laboratory technicians, phlebotomists)
* Students who have previously experience in interprofessional learning activities
* Students who have previously experience in the simulation center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Knowledge and Practices during the simulation | 10 minutes - During the simulation scenarios
  Purposefully Developed 6-item Checklist

SECONDARY OUTCOMES:
General Self Efficacy Scale - GSE | 10 minutes Pre-intervention and post-intervention
  A 10-item questionnaire assessing the level of self-efficacy
Student Satisfaction and Self-Confidence in Learning - SCLS | Post-intervention
  A 13-item questionnaire assessing the self-confidence acquired in learning
Interdisciplinary Education Perception Scale - IEPS | 10 minutes Pre-intervention and post-intervention
  A 18-item questionnaire targeted at evaluating the perception of interprofessional education
Readiness for Interprofessional Learning Scale - RIPLS | 10 minutes Pre-intervention and post-intervention
  A 19-item questionnaire targeted at evaluating the readiness for interprofessional education
Satisfaction with simulation experience - SSE | Post-intervention
  A 18-item questionnaire to assess the perceived satisfaction with simulation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Torino - Department of Clinical and Biological Sciences, Orbassano, Torino, Italy

IPD SHARING:
Plan to Share IPD: No
Due to ethical restrictions. Aggregated data will be available from the responsible upon reasonable request.